CLINICAL TRIAL: NCT07246993
Title: Targeting Neuroplasticity for Persistent Post-Concussive Cognitive Symptoms: A Trial of tDCS and Cognitive Training 3-12 Months Post-mTBI
Brief Title: Targeting Neuroplasticity for Persistent Post-Concussive Cognitive Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2025-34246
Record Dates: First submitted 2025-10-30; First posted 2025-11-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Persistent Post Concussion Syndrome; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, sham-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active tDCS + Cognitive Training (Active Comparator)
  Interventions: Device: Active tDCS
- Sham tDCS + Cognitive Training (Placebo Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — All participants will receive 10 sessions of cognitive training focused on executive functions, delivered over approximately 3 weeks. Cognitive training will be completed on a lab provided computer using PositScience BrainHQ or TaskFlow software. Concurrently, during each training session, participants will receive either active or sham tDCS. Stimulation will be delivered via saline-soaked sponge electrodes using the Soterix 1x1 miniCT TES device. The anode (active electrode) will be placed over the L-DLPFC (approximated by EEG coordinate F3) and the cathode (reference electrode) over the contralateral supraorbital area (Fp2). The active tDCS group will receive 2mA constant current for 20 minutes.
  Arms: Active tDCS + Cognitive Training
Device: Sham tDCS — All participants will receive 10 sessions of cognitive training focused on executive functions, delivered over approximately 3 weeks. Cognitive training will be completed on a lab provided computer using PositScience BrainHQ or TaskFlow software. Concurrently, during each training session, participants will receive either active or sham tDCS. Stimulation will be delivered via saline-soaked sponge electrodes using the Soterix 1x1 miniCT TES device. The anode (active electrode) will be placed over the L-DLPFC (approximated by EEG coordinate F3) and the cathode (reference electrode) over the contralateral supraorbital area (Fp2). The sham tDCS group will receive a brief ramp up and ramp down of current at the beginning and end of the 20 minutes to mimic the sensation of active stimulation.
  Arms: Sham tDCS + Cognitive Training

SUMMARY:
This project investigates an innovative combination of non-invasive neuromodulation (transcranial direct current stimulation - tDCS) and cognitive training as a novel treatment approach aimed at improving function in individuals suffering from persistent post-concussive syndrome (PPCS) following mild traumatic brain injury (mTBI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Has sustained a single mTBI 3-12 months prior to enrollment
* Meets criteria for PPCS (assessed using the CP Screen)
* Has reliable access to a smartphone

Exclusion Criteria:

* Inability to provide informed consent or complete study procedures
* History of moderate/severe TBI
* Significant neurological or psychiatric disorders (other than PPCS-related symptoms like mild depression/anxiety)
* Substance dependence within the last six months
* Contraindications to tDCS (e.g., implanted metal, skin lesions on scalp)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of active tDCS combined with cognitive training compared to sham tDCS combined with cognitive training for improving executive function in individuals with PPCS | Week 4
  Using score on Penn Cognitive Battery

SECONDARY OUTCOMES:
Effects of active versus sham tDCS combined with cognitive training on self-reported affect, stress, cognition, and objectively measured sleep and activity levels | Week 4
  Ecological Momentary Assessment Survey score

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lim, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No